CLINICAL TRIAL: NCT05712590
Title: The Influence of the Nutritional Status of Women Between 30 and 45 Years of Age on the Condition of the Skin and Body Composition
Acronym: VEGOMNI
Status: Completed | Type: Observational
Sponsor: VIST - Faculty of Applied Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: VIST VEGOMNI 11-2022
Record Dates: First submitted 2022-12-07; First posted 2023-02-03 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-04

CONDITIONS: Skin Condition; Body Composition
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Vegans: In this group women aged 30-45 years that follow vegan diet for at least 3 years will be included.
  Interventions: Other: dietary habit
- Vegetarians: In this group women aged 30-45 years that follow vegetarian (lacto-ovo/lacto/ovo) diet for at least 3 years will be included.
  Interventions: Other: dietary habit
- Omnivores: In this group women aged 30-45 years that follow omnivorous diet for at least 3 years will be included.
  Interventions: Other: dietary habit

INTERVENTIONS:
Other: dietary habit — As it is observational study, women that follow three different dietary patterns will be inlcuded .

SUMMARY:
Goal is to investigate the differences in skin condition and body composition among women with different dietary habits aged 30-45 years. Study will be focused onto sub-groups of female subjects following omnivorous, vegetarian or vegan diet.

DETAILED DESCRIPTION:
Investigators will investigate differences among female subjects aged 30-45 years following one of the following diet for at least 3 years:

* vegan
* vegetarian
* omnivorous

Study will focus into the differences in dermal protein density and dermal thickness, skin hydration and trans-epidermal water loss. Study will focus also into body composition, specifically into % of body fat and % of lean body weight.

ELIGIBILITY:
Inclusion Criteria:

* women
* aged 30-45 years
* vegan or vegetarian or omnivorous diet for at least 3 years,
* body mass index (BMI) between 18.5 and 25.

Exclusion Criteria:

* smoking or have smoked in the past (quit less than 3 years ago),
* pregnancy or breastfeeding,
* pre-menopause
* medications that increase skin dryness (e.g. retinoids),
* visiting solariums,
* visiting of the fitness center more than 3 times a week,
* regular consumption of protein supplements (including food supplements with collagen),
* chronic and acute skin diseases,
* chronic and acute diseases of the gastrointestinal tract (e.g. celiac disease),
* lactose intolerance,
* various diets (e.g. health, slimming),
* damaged skin in the test area (inner forearm),
* hyperhidrosis or increased sweating,
* diseases that cause a chronically damaged skin barrier (e.g. atopic dermatitis, ichthyosis),
* cancer diseases,
* pacemaker.

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Healthy women aged 30-45 years following vegan or vegetarian or omnivorous diet for at least 3 years.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Dermal density | baseline
  It will be measured on forearm using ultrasonography as score 0-100.
Dermal thickness | baseline
  It will be measured on forearm using ultrasonography in micrometeres.
Skin hydration | baseline
  It will be measured on forearm using Cortex DermaLab flat hydration probe in microsiemens.
Skin elasticity | baseline
  It will be measured on forearm using Cortex DermaLab elasticity probe in MPa.
Trans epidermal water loss | baseline
  It will be measured on forearm using Cortex DermaLab open-chamberTEWL probe.
% of lean body weight | baseline
  It will be measured using Multiscan is a spectroscopy (BIS).
% of body fat | baseline
  It will be measured using Multiscan is a spectroscopy (BIS).

CONTACTS AND LOCATIONS:
Overall Officials: Katja Žmitek, PhD, Study Director — VIST Higher school of applied sciences
Locations (1):
- VIST - Faculty of applied sciences, Institute of Cosmetics, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No